CLINICAL TRIAL: NCT03535038
Title: Agreement Test of Intravascular Volume Assessment Between Inferior Vena Cava (IVC) Diameter and Vascular Pedicle Width (VPW)
Brief Title: Measurement of Intravascular Volume Using USG of IVC Diameter Compared to VPW Chest X-ray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Amir S Madjid, Anesthesiologist, Indonesia University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IndonesiaUAnes023
Record Dates: First submitted 2018-05-12; First posted 2018-05-24 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Unintubated Patients in ICU and Resuscitation Room
Keywords: Intravascular volume; Inferior vena cava diameter; Ultrasonography; Vascular Pedicle Width; Chest x-ray

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior vena cava (IVC) diameter (Experimental): subjects underwent IVC diameter measurement after VPW measurement
  Interventions: Diagnostic Test: Inferior vena cava (IVC) diameter using USG
- Vascular pedicle width (VPW) (Active Comparator): Supine chest x ray was done and the VPW is assessed by radiologists.
  Interventions: Diagnostic Test: Vascular pedicle width (VPW)

INTERVENTIONS:
Diagnostic Test: Inferior vena cava (IVC) diameter using USG — IVC diameter is measured from the distal of right hepatic pain and inferior vena cava meeting point using Philips En Visor C USG.
  Arms: Inferior vena cava (IVC) diameter
Diagnostic Test: Vascular pedicle width (VPW) — VPW is measured by drawing a line from the left subclavian artery exit point from aorta perpendicular to the point where superior vena cava crosses with right bronchi.
  Arms: Vascular pedicle width (VPW)

SUMMARY:
This study aimed to know the consistency of intravascular volume measurement using USG of IVC compared to VPW chest x-ray

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Validation and reliability test were done for USG operators by assessing IVC in 20 patients supervised by intensivists. Subjects were given informed consent before participating in the study. Subjects underwent the chest x-ray examination with supine position. The measurement of VPW was done by radiologists, considered normal if the value is 53 ± 5 mm, overload if VPW > 71 mm. The subjects then underwent the IVC diameter measurement using USG Philips En Visor C, with transthoracal subcostal approach. The result is considered normal if IVC diameter is 1.5 - 2.5 cm and overload if >2.5 cm, otherwise the subjects is excluded. If the IVC can not be done, subjects will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Adult non-intubated patients aged 18-65 in ICU or resucitation room
* BMI 18.5-35 kg/m2
* Signed informed consent of the patient to be included in the study

Exclusion Criteria:

* BMI >35, intubated
* History of thoracic or heart surgery
* History of external and internal radiation
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Intravascular volume measurement | IVC is measured 30 minutes after VPW
  Measured by VPW and IVC diameter using USG

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beaubien-Souligny W, Bouchard J, Desjardins G, Lamarche Y, Liszkowski M, Robillard P, Denault A. Extracardiac Signs of Fluid Overload in the Critically Ill Cardiac Patient: A Focused Evaluation Using Bedside Ultrasound. Can J Cardiol. 2017 Jan;33(1):88-100. doi: 10.1016/j.cjca.2016.08.012. Epub 2016 Aug 24. PMID 27887762
- [Background] Ferrada P, Anand RJ, Whelan J, Aboutanos MA, Duane T, Malhotra A, Ivatury R. Qualitative assessment of the inferior vena cava: useful tool for the evaluation of fluid status in critically ill patients. Am Surg. 2012 Apr;78(4):468-70. PMID 22472406
- [Background] Cordemans C, De Laet I, Van Regenmortel N, Schoonheydt K, Dits H, Huber W, Malbrain ML. Fluid management in critically ill patients: the role of extravascular lung water, abdominal hypertension, capillary leak, and fluid balance. Ann Intensive Care. 2012 Jul 5;2(Suppl 1 Diagnosis and management of intra-abdominal hyperten):S1. doi: 10.1186/2110-5820-2-S1-S1. eCollection 2012. PMID 22873410
- [Background] Dass B, Shimada M, Kambhampati G, Ejaz NI, Arif AA, Ejaz AA. Fluid balance as an early indicator of acute kidney injury in CV surgery. Clin Nephrol. 2012 Jun;77(6):438-44. doi: 10.5414/cn107278. PMID 22595385
- [Background] Grams ME, Estrella MM, Coresh J, Brower RG, Liu KD; National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome Network. Fluid balance, diuretic use, and mortality in acute kidney injury. Clin J Am Soc Nephrol. 2011 May;6(5):966-73. doi: 10.2215/CJN.08781010. Epub 2011 Mar 10. PMID 21393482
- [Background] Rosenberg AL, Dechert RE, Park PK, Bartlett RH; NIH NHLBI ARDS Network. Review of a large clinical series: association of cumulative fluid balance on outcome in acute lung injury: a retrospective review of the ARDSnet tidal volume study cohort. J Intensive Care Med. 2009 Jan-Feb;24(1):35-46. doi: 10.1177/0885066608329850. Epub 2008 Dec 22. PMID 19103612
- [Background] Stein A, de Souza LV, Belettini CR, Menegazzo WR, Viegas JR, Costa Pereira EM, Eick R, Araujo L, Consolim-Colombo F, Irigoyen MC. Fluid overload and changes in serum creatinine after cardiac surgery: predictors of mortality and longer intensive care stay. A prospective cohort study. Crit Care. 2012 May 31;16(3):R99. doi: 10.1186/cc11368. PMID 22651844
- [Background] Magee G, Zbrozek A. Fluid overload is associated with increases in length of stay and hospital costs: pooled analysis of data from more than 600 US hospitals. Clinicoecon Outcomes Res. 2013 Jun 26;5:289-96. doi: 10.2147/CEOR.S45873. Print 2013. PMID 23836999
- [Background] Wichansawakul S, Vilaichone W, Tongyoo S, Permpikul C, Wonglaksanapimol S, Daengnim K, Suwanboonrit G. Evaluation of correlation between vascular pedicle width and intravascular volume status in Thai critically ill patients. J Med Assoc Thai. 2011 Feb;94 Suppl 1:S181-7. PMID 21721445
- [Background] Kalantari K, Chang JN, Ronco C, Rosner MH. Assessment of intravascular volume status and volume responsiveness in critically ill patients. Kidney Int. 2013 Jun;83(6):1017-28. doi: 10.1038/ki.2012.424. Epub 2013 Jan 9. PMID 23302716
- [Background] Farshidpanah S, Klein W, Matus M, Sai A, Nguyen HB. Validation of the vascular pedicle width as a diagnostic aid in critically ill patients with pulmonary oedema by novice non-radiology physicians-in-training. Anaesth Intensive Care. 2014 May;42(3):321-9. doi: 10.1177/0310057X1404200308. PMID 24794471
- [Background] Nik Muhamad NA, Safferi RS, Robertson CE. Internal Jugular Vein Height and Inferior Vena Cava Diameter Measurement using Ultrasound to Determine Central Venous Pressure: A Correlation Study. Med J Malaysia. 2015 Apr;70(2):63-6. PMID 26162379
- [Background] Miller RR, Ely EW. Radiographic measures of intravascular volume status: the role of vascular pedicle width. Curr Opin Crit Care. 2006 Jun;12(3):255-62. doi: 10.1097/01.ccx.0000224871.31947.8d. PMID 16672786
- [Background] Celebi Yamanoglu NG, Yamanoglu A, Parlak I, Pinar P, Tosun A, Erkuran B, Aydinok G, Torlak F. The role of inferior vena cava diameter in volume status monitoring; the best sonographic measurement method? Am J Emerg Med. 2015 Mar;33(3):433-8. doi: 10.1016/j.ajem.2014.12.014. Epub 2014 Dec 18. PMID 25616587
- [Background] Frank Peacock W, Soto KM. Current technique of fluid status assessment. Congest Heart Fail. 2010 Jul;16 Suppl 1:S45-51. doi: 10.1111/j.1751-7133.2010.00166.x. PMID 20653711
- [Background] Kent A, Patil P, Davila V, Bailey JK, Jones C, Evans DC, Boulger CT, Adkins E, Balakrishnan JM, Valiyaveedan S, Galwankar SC, Bahner DP, Stawicki SP. Sonographic evaluation of intravascular volume status: Can internal jugular or femoral vein collapsibility be used in the absence of IVC visualization? Ann Thorac Med. 2015 Jan-Mar;10(1):44-9. doi: 10.4103/1817-1737.146872. PMID 25593607
- [Background] Salahuddin N, Hussain I, Alsaidi H, Shaikh Q, Joseph M, Hawa H, Maghrabi K. Measurement of the vascular pedicle width predicts fluid repletion: a cross-sectional comparison with inferior vena cava ultrasound and lung comets. J Intensive Care. 2015 Dec 22;3:55. doi: 10.1186/s40560-015-0121-4. eCollection 2015. PMID 26702359
- [Background] Thanakitcharu P, Charoenwut M, Siriwiwatanakul N. Inferior vena cava diameter and collapsibility index: a practical non-invasive evaluation of intravascular fluid volume in critically-ill patients. J Med Assoc Thai. 2013 Mar;96 Suppl 3:S14-22. PMID 23682518
- [Background] Wang H, Shi R, Mahler S, Gaspard J, Gorchynski J, D'Etienne J, Arnold T. Vascular pedicle width on chest radiograph as a measure of volume overload: meta-analysis. West J Emerg Med. 2011 Nov;12(4):426-32. doi: 10.5811/westjem.2011.3.2023. PMID 22224132
- [Background] Marx G, Schindler AW, Mosch C, Albers J, Bauer M, Gnass I, Hobohm C, Janssens U, Kluge S, Kranke P, Maurer T, Merz W, Neugebauer E, Quintel M, Senninger N, Trampisch HJ, Waydhas C, Wildenauer R, Zacharowski K, Eikermann M. Intravascular volume therapy in adults: Guidelines from the Association of the Scientific Medical Societies in Germany. Eur J Anaesthesiol. 2016 Jul;33(7):488-521. doi: 10.1097/EJA.0000000000000447. No abstract available. PMID 27043493
- [Background] Mackenzie DC, Noble VE. Assessing volume status and fluid responsiveness in the emergency department. Clin Exp Emerg Med. 2014 Dec 31;1(2):67-77. doi: 10.15441/ceem.14.040. eCollection 2014 Dec. PMID 27752556
- [Background] Zhang Z, Xu X, Ye S, Xu L. Ultrasonographic measurement of the respiratory variation in the inferior vena cava diameter is predictive of fluid responsiveness in critically ill patients: systematic review and meta-analysis. Ultrasound Med Biol. 2014 May;40(5):845-53. doi: 10.1016/j.ultrasmedbio.2013.12.010. Epub 2014 Feb 2. PMID 24495437
- [Background] Bouchard J, Soroko SB, Chertow GM, Himmelfarb J, Ikizler TA, Paganini EP, Mehta RL; Program to Improve Care in Acute Renal Disease (PICARD) Study Group. Fluid accumulation, survival and recovery of kidney function in critically ill patients with acute kidney injury. Kidney Int. 2009 Aug;76(4):422-7. doi: 10.1038/ki.2009.159. Epub 2009 May 13. PMID 19436332
- [Background] Murphy CV, Schramm GE, Doherty JA, Reichley RM, Gajic O, Afessa B, Micek ST, Kollef MH. The importance of fluid management in acute lung injury secondary to septic shock. Chest. 2009 Jul;136(1):102-109. doi: 10.1378/chest.08-2706. Epub 2009 Mar 24. PMID 19318675
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Lyon M, Blaivas M, Brannam L. Sonographic measurement of the inferior vena cava as a marker of blood loss. Am J Emerg Med. 2005 Jan;23(1):45-50. doi: 10.1016/j.ajem.2004.01.004. PMID 15672337
- [Background] Zhang J, Critchley LA. Inferior Vena Cava Ultrasonography before General Anesthesia Can Predict Hypotension after Induction. Anesthesiology. 2016 Mar;124(3):580-9. doi: 10.1097/ALN.0000000000001002. PMID 26771910
- [Background] Sakurai T, Ando Y, Masunaga Y, Kusano E, Asano Y. Diameter of the inferior vena cava as an index of dry weight in patients undergoing CAPD. Perit Dial Int. 1996 Mar-Apr;16(2):183-5. No abstract available. PMID 9147557
- [Background] Sefidbakht S, Assadsangabi R, Abbasi HR, Nabavizadeh A. Sonographic measurement of the inferior vena cava as a predictor of shock in trauma patients. Emerg Radiol. 2007 Jul;14(3):181-5. doi: 10.1007/s10140-007-0602-4. Epub 2007 Jun 1. PMID 17541661
- [Background] Zengin S, Al B, Genc S, Yildirim C, Ercan S, Dogan M, Altunbas G. Role of inferior vena cava and right ventricular diameter in assessment of volume status: a comparative study: ultrasound and hypovolemia. Am J Emerg Med. 2013 May;31(5):763-7. doi: 10.1016/j.ajem.2012.10.013. Epub 2013 Apr 17. PMID 23602752
- [Background] Brennan JM, Blair JE, Goonewardena S, Ronan A, Shah D, Vasaiwala S, Brooks E, Levy A, Kirkpatrick JN, Spencer KT. A comparison by medicine residents of physical examination versus hand-carried ultrasound for estimation of right atrial pressure. Am J Cardiol. 2007 Jun 1;99(11):1614-6. doi: 10.1016/j.amjcard.2007.01.037. Epub 2007 Apr 18. PMID 17531592
- [Background] Zhao J, Wang G. Inferior Vena Cava Collapsibility Index is a Valuable and Non-Invasive Index for Elevated General Heart End-Diastolic Volume Index Estimation in Septic Shock Patients. Med Sci Monit. 2016 Oct 20;22:3843-3848. doi: 10.12659/msm.897406. PMID 27762259
- [Background] Eisenhuber E, Schaefer-Prokop CM, Prosch H, Schima W. Bedside chest radiography. Respir Care. 2012 Mar;57(3):427-43. doi: 10.4187/respcare.01712. PMID 22391269
- [Background] Ely EW, Haponik EF. Using the chest radiograph to determine intravascular volume status: the role of vascular pedicle width. Chest. 2002 Mar;121(3):942-50. doi: 10.1378/chest.121.3.942. PMID 11888980
- [Background] Taghizadieh A, Nia KS, Moharramzadeh P, Pouraghaei M, Ghavidel A, Parsian Z, Mahmoodpoor A. The PCQP Score for Volume Status of Acutely Ill Patients: Integrating Vascular Pedicle Width, Caval Index, Respiratory Variability of the QRS Complex and R Wave Amplitude. Indian J Crit Care Med. 2017 Nov;21(11):726-732. doi: 10.4103/ijccm.IJCCM_275_17. PMID 29279632
- [Background] Michard F. Underutilized tools for the assessment of intravascular volume status. Chest. 2003 Jul;124(1):414-5; author reply 415-6. No abstract available. PMID 12853559
- [Background] Rice TW, Ware LB, Haponik EF, Chiles C, Wheeler AP, Bernard GR, Steingrub JS, Hite RD, Matthay MA, Wright P, Ely EW; NIH NHLBI ARDS Network. Vascular pedicle width in acute lung injury: correlation with intravascular pressures and ability to discriminate fluid status. Crit Care. 2011;15(2):R86. doi: 10.1186/cc10084. Epub 2011 Mar 7. PMID 21385351
- [Background] Thomason JW, Ely EW, Chiles C, Ferretti G, Freimanis RI, Haponik EF. Appraising pulmonary edema using supine chest roentgenograms in ventilated patients. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1600-8. doi: 10.1164/ajrccm.157.5.9708118. PMID 9603144